CLINICAL TRIAL: NCT06539910
Title: Modified Triple Injection Peri-Sartorius (TIPS) Block for Postoperative Analgesia After Total Knee Arthroplasty (TKA)
Brief Title: Modified TIPS Block for Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, moustafa abdelaziz, Professor of Anaesthesia and Surgical Intensive Care, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0306646
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Knee Arthropathy; Anesthesia, Local
Keywords: Analgesia, arthroplasty, knee replacement, nerve block, peri-sartorial block, triple injection, visual analogue scale
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified TIPS Block (Experimental): Modified Triple Injection Peri-sartorial Block Patients will receive ultrasound guided single puncture triple injections through medial to lateral approach. LA will be injected at the distal FT lateral to the superficial femoral artery (FA), deep to adductor longus muscle (ALM), and at the supra-sartorial plane
  Interventions: Procedure: General Anesthesia; Procedure: TIPS block; Procedure: Mutimodal analgesia
- TIPS Block (Active Comparator): Triple Injection Peri-sartorial Block Patients will receive distal FTB through conventional lateral to medial approach, in addition to a supra-sartorial plane injection
  Interventions: Procedure: General Anesthesia; Procedure: Modified TIPS block; Procedure: Mutimodal analgesia

INTERVENTIONS:
Procedure: General Anesthesia — All blocks will be performed after induction of general anaesthesia (GA). Upon arrival to the operating room (OR), a multichannel monitor will be attached to patients, followed by the administration of 2 mg midazolam IV after securing an IV cannula. Controlled GA via a laryngeal mask airway (LMA) will be done to all patients
Procedure: TIPS block — Patients will receive distal FTB through conventional lateral to medial approach, in addition to a supra-sartorial plane injection. Distal adductor canal block via another needle puncture.Ten mL of a mixture of 0.25 % bupivacaine and 8 mg dexamethasone will be injected in the suprasartorial plane and 20 mL will be injected at the distal adductor canal.Ten mL of the LA mixture will be injected 2 cm above the FT apex via ultrasound guided in-plane lateral to medial approach just lateral to the superficial femoral artery
  Arms: Modified TIPS Block
Procedure: Modified TIPS block — Patients will receive ultrasound guided single puncture triple injections through medial to lateral approach. LA will be injected at the distal FT lateral to the superficial femoral artery (FA), deep to adductor longus muscle (ALM), and at the supra-sartorial plane.Both groups will receive a mixture of 0.25 % bupivacaine and 8 mg dexamethasone. Ten mL will be injected in the suprasartorial plane and 20 mL will be injected at the distal adductor canal.Ten mL of the LA anaesthetic mixture will be injected 2 cm above the FT apex via ultrasound guided in-plane medial to lateral approach just lateral to the superficial femoral artery. Then, the needle will be redirected just underneath the ALM and 10 mL of the LA mixture will be injected in the plane between the ALM and the adductor magnus muscle (AMM).Total volume of LA will be 50 mL.
  Arms: TIPS Block
Procedure: Mutimodal analgesia — Postoperatively, multimodal analgesia regimen will be continued in the form of paracetamol 1 g /8 hours and ketorolac 30 mg /8 hours intravenously for 24 hours. Intravenous morphine patient controlled analgesia will be started at the end of surgery at a concentration of 0.5 mg/ml without a background infusion on a demand dose of 1 mg with a lockout interval of 10 minutes

SUMMARY:
The is carried out to compare triple injection peri-sartorial block to a modified block including an extra local anesthetic injection deep to the adductor longs muscle via a medial to lateral approach regarding the peri-operative analgesia following total knee arthroplasty (TKA)

DETAILED DESCRIPTION:
We hypothesise that LA injection at a plane deep to adductor longus muscle at the level of femoral triangle may block the 2 divisions of the ON and improve analgesia following TKA. Moreover, the medial to lateral needle trajectory may avoid NVM injury.

Aim of the work: The primary aim of this study is to determine if addition of LA injection underneath the ALM targeting ON divisions to tri-injection perisartorius (TIPS) block, may decrease the postoperative opioid rescue analgesic requirements after TKA.

The secondary aim of this study is to investigate the effect of addition of LA injection under the ALM to TIPS block on the resting and dynamic VAS scores during the 1st 24 h postoperative period. The secondary aims include the time to the 1st request of rescue analgesia, the motor power of the operated limb as well as any complication related to the block technique.

Methods: After obtaining approval from Alexandria university ethics committee, this study will be carried out in El-Hadara university hospital on American Society of Anesthesiologists (ASA) physical status I-III 90 patients scheduled for unilateral TKA. Based on a pilot study, a total sample size of 90 participants - 45 patients in TIPS group and 45 patients in mTIPS group - is needed to achieve 80% power and to detect difference of 0.6 mg in the mean of morphine consumption between the two groups with group standard deviations of 1 Using t test (a two-sided two-sample t-test) at a significance level of 05. Sample size was calculated using NCSS 2004 and PASS 2000 program. Informed written consent will be signed by all patients. The visual analogue scale (VAS) score interpretation and the use of patient controlled analgesia (PCA) device will be explained to all participants. The exclusion criteria will include; BMI > 35 kg/m2, pre-existing neurological deficit, any disability of the non-operated limb preventing fair mobilization, known contraindications to peripheral nerve block (coagulopathy or infection at the site of injection), or chronic opioid users/abusers. Patients will be randomised into 2 groups using a closed envelope technique:

Group TIPS: patients will receive distal FTB through conventional lateral to medial approach, in addition to a supra-sartorial plane injection.

Group MTIPS: patients will receive ultrasound guided single puncture triple injections through medial to lateral approach. LA will be injected at the distal FT lateral to the superficial femoral artery (FA), deep to adductor longus muscle (ALM), and at the supra-sartorial plane.

Both groups will receive distal adductor canal block via another needle puncture.

All blocks will be performed after induction of general anaesthesia (GA). Upon arrival to the operating room (OR), a multichannel monitor will be attached to patients, followed by the administration of 2 mg midazolam IV after securing an IV cannula. Controlled GA via a laryngeal mask airway (LMA) will be done to all patients

Both groups will receive a mixture of 0.25 % bupivacaine and 8 mg dexamethasone. Ten mL will be injected in the suprasartorial plane and 20 mL will be injected at the distal adductor canal. The total volume of LA will be determined according to group selection:

Group TIPS: Ten mL of the LA mixture will be injected 2 cm above the FT apex via ultrasound guided in-plane lateral to medial approach just lateral to the superficial femoral artery. Then, the needle will be redirected to perform the suprasartorial plane injection. Total volume of LA will be 40 mL.

Group MTIPS: Ten mL of the LA anaesthetic mixture will be injected 2 cm above the FT apex via ultrasound guided in-plane medial to lateral approach just lateral to the superficial femoral artery. Then, the needle will be redirected just underneath the ALM and 10 mL of the LA mixture will be injected in the plane between the ALM and the adductor magnus muscle (AMM). Again, the needle will be redirected to perform the suprasartorial plane injection. Total volume of LA will be 50 mL.

Postoperatively, multimodal analgesia regimen will be continued in the form of paracetamol 1 g /8 hours and ketorolac 30 mg /8 hours intravenously for 24 hours. Intravenous morphine patient controlled analgesia will be started at the end of surgery at a concentration of 0.5 mg/ml without a background infusion on a demand dose of 1 mg with a lockout interval of 10 minutes. The time to the 1st demand dose of rescue analgesia will be recorded. Resting and dynamic VAS assessment will be carried out every 4 hours during the 24 h follow up period. Total postoperative morphine requirements will be measured during the 24 h postoperative follow up period. Postoperative functional outcome will be assessed using the Timed Up and Go (TUG) test and the 30-second Chair Stand Test (30s-CST) in the evening of the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* BMI > 35 kg/m2 Pre-existing neurological deficit Any disability of the non-operated limb preventing fair mobilization Known contraindications to peripheral nerve block (coagulopathy or infection at the site of injection) Chronic opioid users/abusers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid rescue analgesic requirements | 24 hours
  Intravenous morphine patient controlled analgesia will be started at the end of surgery at a concentration of 0.5 mg/ml without a background infusion on a demand dose of 1 mg with a lockout interval of 10 minutes. Total postoperative morphine consumption will be measured

SECONDARY OUTCOMES:
The time to the 1st demand dose of rescue analgesia | 24 hours
  The time to the 1st demand dose of rescue analgesia will be recorded
Resting and dynamic VAS assessment | 24 hours
  Resting and dynamic VAS assessment will be carried out every 4 hours
Timed Up and Go (TUG) test | 24 hours
  Timed Up and Go (TUG) test
30-second Chair Stand Test (30s-CST) | 24 hours
  30-second Chair Stand Test (30s-CST)

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request via mail to the principal investigator

REFERENCES:
- [Result] Woodworth GE, Arner A, Nelsen S, Nada E, Elkassabany NM. Pro and Con: How Important Is the Exact Location of Adductor Canal and Femoral Triangle Blocks? Anesth Analg. 2023 Mar 1;136(3):458-469. doi: 10.1213/ANE.0000000000006234. Epub 2023 Feb 17. PMID 36806233